CLINICAL TRIAL: NCT04353310
Title: Evaluating the Effects of Curcumin in Moderate to Severe Asthmatics
Brief Title: Evaluating Effects of Curcumin in Moderate to Severe Asthmatics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5190424; 145101 (Other: FDA)
Record Dates: First submitted 2019-11-13; First posted 2020-04-20 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: asthma; curcumin
MeSH Terms: conditions — Asthma | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental)
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Curcumin 1500mg PO BID
  Arms: Curcumin
Other: Placebo — identical in appearance to curcumin
  Arms: Placebo

SUMMARY:
The purpose of this investigator-initiated study is to evaluate the effects of oral curcumin supplementation versus placebo in adult patients with moderate to severe asthma. Curcumin, a derivative of turmeric, has been shown in animal models to inhibit the secretion of pro-inflammatory cytokines and decrease airway constriction and hyperreactivity with only a few observational studies available in humans with discordant results.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 and older
4. Physician diagnosed moderate to severe asthma: (GINA 2018)

   a. Stable asthma that requires ICS/LABA and/or an additional controller agent (i.e. LTRA, LAMA)
5. Ability to take oral medication and be willing to adhere to the regimen
6. Ability to speak and read English
7. If female and sexually active, should use effective forms of birth control

Exclusion Criteria:

1. Current use of turmeric (curcumin) or use within the last 7 days
2. Current use of biologic therapy/ immunotherapy/ or bronchothermoplasty
3. Pregnancy or lactation
4. Known allergic reactions to components of turmeric (curcumin)
5. Current use of anticoagulants, and history of coagulopathy or liver disease
6. INR greater than 2.0, PTT greater than 45.0 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Asthma Control | 3 months
  defined by the Asthma Control Test, which has a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled)

SECONDARY OUTCOMES:
Number of Severe Asthma Exacerbations in 3 Months | 3 months
Cumulative Days Missed From School or Work in 3 Months | 3 months
Spirometry | 3 months
  FEV1/FVC ratio, FEV1: forced expiratory volume in one second, FVC: forced vital capacity
Exhaled nitric oxide | 3 months
Total IgE | 3 months
Total plasma eosinophil count | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laren Tan, MD, Principal Investigator — Loma Linda University Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Szefler SJ, Sullivan SD, Thomas MD, Wenzel SE, Reddel HK. A new perspective on concepts of asthma severity and control. Eur Respir J. 2008 Sep;32(3):545-54. doi: 10.1183/09031936.00155307. PMID 18757695
- [Background] Aggarwal BB, Surh YJ, Shishodia S (Eds.). Mol. Targets Ther. Uses Curcumin Health Dis, Springer, US. 2007; 1-75.
- [Background] Baldwin AS Jr. Series introduction: the transcription factor NF-kappaB and human disease. J Clin Invest. 2001 Jan;107(1):3-6. doi: 10.1172/JCI11891. No abstract available. PMID 11134170
- [Background] Oh SW, Cha JY, Jung JE, Chang BC, Kwon HJ, Lee BR, Kim DY. Curcumin attenuates allergic airway inflammation and hyper-responsiveness in mice through NF-kappaB inhibition. J Ethnopharmacol. 2011 Jul 14;136(3):414-21. doi: 10.1016/j.jep.2010.07.026. Epub 2010 Jul 17. PMID 20643202
- [Background] Liu L, Shang Y, Li M, Han X, Wang J, Wang J. Curcumin ameliorates asthmatic airway inflammation by activating nuclear factor-E2-related factor 2/haem oxygenase (HO)-1 signalling pathway. Clin Exp Pharmacol Physiol. 2015 May;42(5):520-9. doi: 10.1111/1440-1681.12384. PMID 25739561
- [Background] Wong CK, Li ML, Wang CB, Ip WK, Tian YP, Lam CW. House dust mite allergen Der p 1 elevates the release of inflammatory cytokines and expression of adhesion molecules in co-culture of human eosinophils and bronchial epithelial cells. Int Immunol. 2006 Aug;18(8):1327-35. doi: 10.1093/intimm/dxl065. Epub 2006 Jun 23. PMID 16798840
- [Background] Wuyts WA, Vanaudenaerde BM, Dupont LJ, Demedts MG, Verleden GM. Involvement of p38 MAPK, JNK, p42/p44 ERK and NF-kappaB in IL-1beta-induced chemokine release in human airway smooth muscle cells. Respir Med. 2003 Jul;97(7):811-7. doi: 10.1016/s0954-6111(03)00036-2. PMID 12854631
- [Background] Kobayashi T, Hashimoto S, Horie T. Curcumin inhibition of Dermatophagoides farinea-induced interleukin-5 (IL-5) and granulocyte macrophage-colony stimulating factor (GM-CSF) production by lymphocytes from bronchial asthmatics. Biochem Pharmacol. 1997 Oct 1;54(7):819-24. doi: 10.1016/s0006-2952(97)00220-7. PMID 9353136
- [Background] Ram A, Das M, Ghosh B. Curcumin attenuates allergen-induced airway hyperresponsiveness in sensitized guinea pigs. Biol Pharm Bull. 2003 Jul;26(7):1021-4. doi: 10.1248/bpb.26.1021. PMID 12843631
- [Background] Kim DH, Phillips JF, Lockey RF. Oral curcumin supplementation in patients with atopic asthma. Allergy Rhinol (Providence). 2011 Apr;2(2):e51-3. doi: 10.2500/ar.2011.2.0016. PMID 22852117
- [Background] Abidi A, Gupta S, Agarwal M, Bhalla HL, Saluja M. Evaluation of Efficacy of Curcumin as an Add-on therapy in Patients of Bronchial Asthma. J Clin Diagn Res. 2014 Aug;8(8):HC19-24. doi: 10.7860/JCDR/2014/9273.4705. Epub 2014 Aug 20. PMID 25302215
- [Background] Gupta SC, Patchva S, Aggarwal BB. Therapeutic roles of curcumin: lessons learned from clinical trials. AAPS J. 2013 Jan;15(1):195-218. doi: 10.1208/s12248-012-9432-8. Epub 2012 Nov 10. PMID 23143785
- [Background] Basnet P, Skalko-Basnet N. Curcumin: an anti-inflammatory molecule from a curry spice on the path to cancer treatment. Molecules. 2011 Jun 3;16(6):4567-98. doi: 10.3390/molecules16064567. PMID 21642934
- [Background] Cheng AL, Hsu CH, Lin JK, Hsu MM, Ho YF, Shen TS, Ko JY, Lin JT, Lin BR, Ming-Shiang W, Yu HS, Jee SH, Chen GS, Chen TM, Chen CA, Lai MK, Pu YS, Pan MH, Wang YJ, Tsai CC, Hsieh CY. Phase I clinical trial of curcumin, a chemopreventive agent, in patients with high-risk or pre-malignant lesions. Anticancer Res. 2001 Jul-Aug;21(4B):2895-900. PMID 11712783
- [Background] Lao CD, Ruffin MT 4th, Normolle D, Heath DD, Murray SI, Bailey JM, Boggs ME, Crowell J, Rock CL, Brenner DE. Dose escalation of a curcuminoid formulation. BMC Complement Altern Med. 2006 Mar 17;6:10. doi: 10.1186/1472-6882-6-10. PMID 16545122
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Derived] Quan M, Alismail A, Daher N, Cleland D, Chavan S, Tan LD. Randomized, placebo controlled, double blinded pilot superiority phase 2 trial to evaluate the effect of curcumin in moderate to severe asthmatics. BMC Pulm Med. 2021 Aug 17;21(1):268. doi: 10.1186/s12890-021-01619-y. PMID 34404358